CLINICAL TRIAL: NCT05285020
Title: Influence of Antigravity Treadmill With Alter G on the Postural Stability of Patients With Traumatic Lower Limb Injuries
Brief Title: Antigravity Treadmill With Alter G on the Postural Stability of Traumatic Lower Limb Injuries
Acronym: ALTERG20
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: FREMAP Mutual Insurance Company for Occupational Accidents and Diseases (Industry)
Responsible Party: Principal Investigator, Esther Melero Baez, Principal Investigator, FREMAP Mutual Insurance Company for Occupational Accidents and Diseases
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CTS954.EM1
Record Dates: First submitted 2021-11-07; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Injury Traumatic; Muscle Injury; Bone Injuries Joints; Tendon Injuries; Lower Limb Injury; Ligament Injury
Keywords: postural balance; lower limb; exercise therapy; rehabilitation; gait; body weight; injury traumatic
MeSH Terms: conditions — Wounds and Injuries; Tendon Injuries; Leg Injuries; Body Weight | interventions — Weights and Measures

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alter G group (Experimental): This group will perform the hospital's standard protocol for these injuries once a day during two weeks.
  They carried out the re-education of the gait (at the parallel bars) with a progressive load in scale controlled by the patient.
  Also, they carried out a re-education of the gait and progressive loading in the system Alter G (anti-gravity treadmill).
  Interventions: Other: Alter G; Other: Parallel bars and Scale; Other: Standard rehabilitation protocol
- Control group (Other): This group will perform the hospital's standard protocol for these injuries once a day during two weeks.
  They just carried out the re-education of the gait (at the parallel bars) with a progressive load in scale controlled by the patient.
  Interventions: Other: Parallel bars and Scale; Other: Standard rehabilitation protocol

INTERVENTIONS:
Other: Alter G — It is anti-gravity treadmill treatment on Alter G. They will start with a 30-50% body weight load during the first week that will be progressively increased to 50-70% during the second (5% more each day during the 10 sessions as far as possible).
  The slope will be 0% and the speed 2-3km/h the first week and 3-4 km/h the second. Treatment will be performed during 15 minutes for two weeks (10 sessions).
  Arms: Alter G group
Other: Parallel bars and Scale — It is a re-education of the gait at the parallel bars with a progressive load in scale controlled by the patient during 10 minutes for two weeks.
Other: Standard rehabilitation protocol — It is the hospital's standard protocol for that injuries once a day for two weeks.

SUMMARY:
This prospective randomised study aimed to test the investigators's hypothesis that anti-gravity treadmill therapy has beneficial effects on postural stability tests over a standard rehabilitation protocol in patients who have suffered traumatic injuries of the lower limb, demonstrating an improvement in the Biodex platform's values.

The total of 30 patients participated in this study (n=30). There were 15 subjects in control group and 15 in experimental group.

DETAILED DESCRIPTION:
This prospective, randomised, controlled, longitudinal and triple-blind masked clinical design was performed in patients derived to the rehabilitation service of Fremap Sevilla Hospital after an laboral accident with surgery and not surgery traumatic injuries.

After that, participants were questioned about their personal data and the inclusion and exclusion criteria. All agreed to participate and provided signed informed consent prior to data collection.

Participants were allocated according to the inclusion and exclusion criteria into an intervention and a control group. The intervention was performed in two weeks. Patients were randomised into the intervention (anti-gravity treadmill) or control (standard protocol) rehabilitation group.

Previous data is taken from the "Postural Stability", "Stability Limits" and " m-CTSIB" tests on the Biodex Balance System SD platform.

The control group will perform the hospital's standard protocol for these injuries while the experimental group will also be added the anti-gravity treadmill in Alter G once a day.

At 2 week post-treatment, subjects were tested again. All patients were able to complete all rehabilitation sessions and balance tests.

Sample size assessment: accepting an alpha risk of 0.05 and a beta risk of 0.1 in a bilateral contrast, 15 subjects in each group are needed to detect a minimum difference of 15% between two groups, assuming that there are 2 groups and a standard deviation of 12%. A 10% rate of loss of insurance has been estimated.

Statistical analysis plan: the statistical analysis will be carried out using IBM-SPSS Statistics 24 software. The Kolmogorov-Smirnov test will be applied to test the distribution of the data. Student's t-test will be applied for paired variables when the data have a parametric distribution. The Mann-Whitney U test will be used to analyse data with a non-parametric distribution. The Chi-Squared will be used to compared qualitative variables. The confidence level used will be 95% (0.05) and the power of the study will be 90% (0.1).

ELIGIBILITY:
Inclusion Criteria:

* Age between 25 and 55
* Sex male and female
* Surgical or non-surgical subacute knee, ankle, and foot traumatic injuries

Exclusion Criteria:

* Vestibular pathology
* Important dysmetry
* Neurological pathology
* Acute inflammatory diseases.
* Important degenerative diseases.
* Autoimmune diseases.
* Severe visual deficits.
* Tumor pathology.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-07-10 (Estimated); Study Completion 2022-07-24 (Estimated)

PRIMARY OUTCOMES:
Postural Stability test | Two weeks
  The Postural Stability Test emphasizes a patient's ability to maintain center of balance. The patient's score on this test assesses deviations from center, thus a lower score is more desirable than a higher score.
LOS test | Two weeks
  This test challenges patients to move and control their center of gravity within their base of sup- port. During each test trial, patients must shift their weight to move the cursor from the center target to a blinking target and back as quickly and with as little deviation as possible. The same process is repeated for each of nine targets. Targets on the screen blink in random order.
m-CTSIB test | Two weeks
  This test provides an assessment of a patient's ability to integrate multiple senses with respect to balance and compensate when one or more of these senses are engaged. This test will be performed under 4 different conditions. It will be carried out bilaterally, first with the static platform and then with the unstable rubber surface to increase the difficulty.

IPD SHARING:
Plan to Share IPD: No